CLINICAL TRIAL: NCT04756661
Title: Carbetocin Versus Combined Oxytocin and Misoprostol for Prevention of Postpartum Hemorrhage in Women With Severe Preeclampsia
Brief Title: Uterotonics for Severe Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CARBOXMISO
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Preeclampsia Severe
MeSH Terms: interventions — carbetocin; Oxytocin; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin (Experimental): Patient received 100 mcg of carbetocin intravenous over one minute immediately after delivery of the baby.
  Interventions: Drug: Carbetocin
- Oxytocin plus misoprostol (Active Comparator): Patient received 10 units of oxytocin IV drip and 400 mcg of misoprostol rectally after anesthesia.
  Interventions: Drug: Oxytocin; Drug: Misoprostol

INTERVENTIONS:
Drug: Carbetocin — 100 mcg of Carbetocin intravenous injection
  Arms: Carbetocin
Drug: Oxytocin — 10 IU oxytocin IV drip
  Arms: Oxytocin plus misoprostol
Drug: Misoprostol — 400 mcg rectal
  Arms: Oxytocin plus misoprostol

SUMMARY:
The study compares the effect of Intravenous carbetocin versus combined use of intravenous oxytocin and rectal misoprostol for prevention of postpartum hemorrhage during delivery of women with severe preeclampsia

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women which diagnosed with severe pre-eclampsia.
* Singleton pregnancy.
* Termination of pregnancy by Cesarean section after 28 weeks of gestation.

Exclusion Criteria:

* Suspected or proven placental abruption.
* Known placenta Previa or acreata.
* Multiple pregnancies.
* Obesity (BMI >35).
* Anemia (<9 g/dl).
* Retained placental tissues.
* Big baby (> 4 kg).
* Presence of coagulopathy.
* Polyhydramnios.
* Presence of Uterine fibroids.
* Medical diseases as; cardiac, liver, renal or endocrine diseases.
* General anesthesia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
The rate of postpartum hemorrhage more than 1000 ml | 30 minutes
  the amount of bleeding during and after CS

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No